CLINICAL TRIAL: NCT04061382
Title: Serum Testing of Representative Youngsters: Sero- Epidemiological Survey of England in 2019/2020
Brief Title: Sero-epidemiological Survey of England in 2019/2020 - COVID-19
Acronym: STORY
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: ID 263097
Record Dates: First submitted 2019-07-30; First posted 2019-08-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Serogroup C Meningococcal Meningitis; Diphtheria; COVID-19
MeSH Terms: conditions — Meningitis, Meningococcal; Diphtheria; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be centrifuged, separated and frozen at local sites at -80°C. Ideally this will happen within 24h with a window of up to 72h. Up to two 2ml aliquots per participant will be shipped to PHE in batches of up to 500 on dry ice. Residual sera beyond this volume will be shipped to the Oxford Vaccine Group(OVG) for storage. For participants where consent is obtained for DNA extraction and storage in the Oxford Vaccine Centre biobank residual blood clots will be shipped to the OVG for this purpose. Participant or their parents will take the oral fluid swab on the day of the visit. Once received by the study team it will be kept in a cool bag until the samples arrive in the lab. They will then be frozen to -80° before being shipped to PHE. Blood samples collected for T cell testing will be shipped to the OVG lab for same-day processing for separation of PBMCs. Saliva samples with be processed in line with local SOPs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Randomised selection of population - Group 1: Group 1 will be focusing on COVID-19, diphtheria and group C invasive meningococcal disease. The investigators are aiming to recruit around 2300 individuals and the investigators are aiming to ensure that sample is broadly representative of the region according to IMD (Index of Multiple Deprivation scores). PHE have generated a list of all postcodes in recruiting regions and determining the quintiles of IMD within that region. Participants interested in taking part in the study will contact sites to arrange a visit. Basic demographic characteristics will be collected by questionnaire and/ or case report form (CRF) and will include: DOB, gender, GP details, Ethnic group, association with communities of special interest, household income and vaccination history.The questionnaire will gather information regarding potential COVID-19 symptoms both in the participant and the participant's household.
  Interventions: Procedure: Venepuncture; Procedure: Oral fluid swab
- Group 2: Group two will focus on 0-19 year olds only. They will not be restricted to the post code sampling. Instead this will include standard recruitment methods such as social media advertisements within the normal recruiting regions for each site. Other methods of recruitment are identification of potential participants by the local study team, staff communication channels and inpatients or outpatients clinics as long as potential participants are not patients. The questionnaire will gather information regarding potential COVID-19 symptoms both in the participant and the participant's household.
  A proportion of participants from this group from selected sites will also provide up to a maximum of three blood samples for separation of peripheral blood mononuclear cells (PBMCs) to evaluate T cell responses. These participants can be either seronegative or seropositive at their Visit 1.
  Interventions: Procedure: Venepuncture; Procedure: Oral fluid swab
- Group 3: Group three will consist of up to 300 participants aged 0-19 from the Black, Asian and Minority ethnic population aged 0-19 years. They will not be restricted to the post code sampling and will be recruited at a sub-set of sites depending on capacity and the demographic profile of the local population. Recruitment will be by multiple approaches, including mail outs, radio and advertising in community (e.g. community centres, religious establishments) or Pharmacies and GP practices where we have ethics approval for them to act as PICs. These can vary according to each site's experience and their contacts within their local community on how is best to approach the BAME community. Other methods of recruitment are identification of potential participants by the local study team, staff communication channels and inpatients or outpatients clinics as long as potential participants are not patients.
  Interventions: Procedure: Venepuncture; Procedure: Oral fluid swab

INTERVENTIONS:
Procedure: Venepuncture — One study visit will be conducted by research study staff and blood sampling will be carried out.
  Up to three follow-up visits will be conducted for a percentage of participants, where additional blood samples will be collected. The blood sample will initially focus on looking at population immunity to diphtheria, group C invasive meningococcal disease and SARS-CoV-2.
Procedure: Oral fluid swab — Saliva sampling will be collected during the follow-up visits. This swab will be collected either by the participant or the participants parent/guardian on the day of the visit. The saliva sampling will primarily be analysed for SARS-CoV-2 antibodies.

SUMMARY:
This is a pilot study to assess the feasibility of establishing a national sero-epidemiological survey in England in individuals aged 0-24 years, focusing on assessing humoral immunity against diphtheria, Group C invasive meningococcus and SARS-CoV-2. The investigators will recruit 2800 to 3800 individuals, divided into three groups:

Group one (N= 2300):

This will include all age groups (0-24years), with recruitment restricted by postcodes provided by Public Health England (PHE) to recruit a representative population for the region as assessed by the IMD (Index of Multiple Deprivation scores).

Group two (N= up to 1200):

This group has been added following additional funding to enhance the sample size in response to the COVID-19 pandemic. This will recruit 0-19 year olds and will not be restricted by post code sampling. Instead recruitment will be by public promotion within the normal recruiting regions for each site.

Group three (N= up to 300):

Addition of Group 3 which is enhanced surveillance in participants from Black, Asian or minority ethnic groups (BAME). Since the start of recruitment we have noted that only 11% of participants are from BAME population, despite recruiting in ethnically diverse regions. Given the increased risk of COVID-19 disease in the BAME community, this is a potential limitation of the study as it stands, not only because it may not reflect the diversity of the UK population, but because it does not allow assessment of whether the differing disease rates and seropositivity in adults are reflected in differences in seropositivity rates in children. Similarly to Group 2, this will recruit 0-19 year olds and will not be restricted by post code sampling.

DETAILED DESCRIPTION:
Public Health England has an ongoing sero-prevalence programme to assess how well the population is protected from vaccine preventable diseases. The current way to check this is by testing left over blood samples from participating healthcare laboratories around the country. However, these samples may not be representative of the general population, particularly in younger age groups who are often most at risk from vaccine preventable diseases. In the Netherlands, they use a different system to assess how well the population is protected from vaccine preventable diseases, actively collecting blood samples from a representative cross section of society. This type of approach would address the limitations of using residual serum samples and allows the collection of additional relevant history e.g. number of family members and previous vaccines received. The investigators are therefore proposing a pilot study to assess the feasibility of establishing a national sero- epidemiological survey in England in individuals aged 0 - 24 years. The investigators will be focusing initially on diphtheria and group C invasive meningococcal disease, both of which are vaccine preventable. This will involve enrolling 2300 participants in the study from different geographical and socioeconomic backgrounds across our test sites and taking a blood sample. This blood will be analysed to look at the level of immunity to vaccine preventable diseases.

The original protocol has been amended to include the testing of antibodies against other infectious diseases, specifically COVID-19. A second group has been added to recruit an additional 500 to 1200 participants between the ages of 0-19 years. The additional funding has been used to open two more sites to recruit to group two across regions on England that are currently not represented by this study. Having a large number of blood samples from a range of age groups is useful when gathering information about an emerging disease such as the current novel coronavirus (COVID-19). These samples can help provide answers regarding the true number of infections with SARS-CoV-2 (the virus which causes COVID-19 disease) in this population. Group 2 can be enhanced by the samples received from other ethically approved research projects where participants have consented for their samples being used outside of the study.

Additional funding has been granted for the addition of 300 participants from the BAME community, who will form Group 3. Data from Group 3 would be invaluable in understanding whether higher rates of disease in the BAME community are a result of greater exposure to COVID-19 contact, a higher likelihood of being infected once exposed or a greater risk of disease once infection occurs.

In addition to increasing the sample size and the number of regions in the UK that are being sampled, a longitudinal sampling cohort has been introduced. A subset of participants equally distributed over the age bands will be enrolled into the longitudinal aspect of the study where repeat blood and saliva samples are taken to look for antibodies against SARS-CoV-2. A questionnaire to ascertain whether the participant or any household contacts have had any symptoms of or been tested positive for COVID-19 will also be collected.

A proportion of participants from this group from selected sites will also provide up to a maximum of three blood samples for separation of peripheral blood mononuclear cells (PBMCs) to evaluate T cell responses. These participants can be either seronegative or seropositive at their Visit 1.

With the latter addition of four more sites, all NHS regions are now represented in the study.

ELIGIBILITY:
Inclusion Criteria:

* Parents/legal guardians or adult participant* is willing and able to give informed consent for participation in the study.
* Male or Female, aged 0 - 24 years inclusive (Group 1)
* Male or Female, aged 0 - 19 years inclusive (Group 2)
* Male or Female, aged 0 - 19 years inclusive with BAME background (Group 3)
* Parents/legal guardians or adult participants are willing to allow their General Practitioner or relevant NHS databases to be contacted for a full immunisation history

Exclusion Criteria:

* If participants do not live in the postcode districts selected by PHE (Group 1 only)
* If participants are not from the BAME population (Group 3 only
* Medically diagnosed bleeding disorder
* Medically diagnosed platelet disorder
* Anticoagulation medication
* Pregnancy
* If another member of their household is participating who is within 5 years of age of the potential participants age

Temporary exclusion criteria:

The participant may not enter the study if they or any member of their household is under temporary isolation measures for suspected SARS-CoV-2 infection.

Ages: 1 Day to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Basic demographic characteristics will be collected by questionnaire and/or case report form (CRF) and will include: DOB, gender, GP details, ethnic group, association with communities of special interest (e.g. faith communities) household income and vaccination history.
  Vaccination history will be verified during serum sample collection using the Red Book or other vaccination records, or checking with the general practitioner or the Child Health Immunisation Service (CHIS) database. Where possible this will include batch information for diphtheria pre-school booster to determine which specific product was received.
Sampling Method: Probability Sample
Enrollment: 2963 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Feasibility of developing an England based sero-epidemiological programme in 0-24 year olds | 11months
  Measure the representativeness of participants as compared to the census data for the study region.
Feasibility of developing an England based sero epidemiological survey in 0-24 year olds | 11 months
  Test serological markers of immunity for vaccine preventable diseases starting with diphtheria.
Feasibility of developing an England based sero epidemiological survey in 0-24 year olds | 11 months
  Test serological markers of immunity for vaccine preventable diseases including Invasive Meningococcal type C.
Feasibility of developing an England based sero epidemiological survey in 0-24 year olds | 11 months
  Test serological markers to determine the true number of infections with SARS-CoV-2 in the population.

SECONDARY OUTCOMES:
Recruitment rate | 11 Months
  Recruitment rate per month, recruitment rates as percentage of potential participants contacted
Cost | 12 months
  Cost per sample obtained of 'disease specific correlates of protection/markers of immunity, e.g. Anti-Diphtheria Toxoid IgG concentrations and Capsular Group C meningococcal Serum bactericidal activity (SBA) titres and Serum IgG to SARS-CoV-2 antigens, including spike and nucleocapsid protein (as measured by ELISA and/or neutralising assay)
To assess, in relevant age groups and different ethnicities antibody concentrations against infections and vaccine preventable diseases | 11 months
  IgG to COVID-19 spike and nucleocapsid protein
Sera collection | 11 months
  * A collection of anonymised sera from participants with appropriate consent and known demographic details and immunisation history.
  * Serum IgG to SARS-CoV-2 antigens, including spike and nucleocapsid protein (as measured by ELISA and/or neutralising assay)
Exploratory | 11 months
  • Representativeness of participants sampled, in terms of the local population's ethnicity, community identity, migrant population and socioeconomic background between groups.
  Differences in immunological read outs
  * PCR for SARS-CoV-2 on saliva samples this will be stored and processed at the end of the study.
  * IgA to SARS-CoV-2 in saliva paired with serum samples.
Exploratory | 6 months
  • T cell responses to SARS-CoV-2 antigens including, but not limited to S, M and N proteins, as measured by techniques including, but not limited to
  * ELISpot
  * ICS
  * Proliferation assay
Exploratory | 6 months
  • Antigen specific IgG and T cells against non-SARS-CoV-2 coronaviruses (e.g. NL62 and 229E)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Snape, Professor, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology & Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ratcliffe H, Tiley KS, Andrews N, Amirthalingam G, Vichos I, Morey E, Douglas NL, Marinou S, Plested E, Aley P, Galiza EP, Faust SN, Hughes S, Murray CS, Roderick M, Shackley F, Oddie SJ, Lees T, Turner DPJ, Raman M, Owens S, Turner P, Cockerill H, Lopez Bernal J, Linley E, Borrow R, Brown K, Ramsay ME, Voysey M, Snape MD. Community seroprevalence of SARS-CoV-2 in children and adolescents in England, 2019-2021. Arch Dis Child. 2023 Jan 19;108(2):123-130. doi: 10.1136/archdischild-2022-324375. PMID 35858775